CLINICAL TRIAL: NCT06533683
Title: Effects of Kinesio Taping Versus Extracorporeal Shock Wave Therapy on Pain in the Treatment of Calcaneal Spur: A Retrospective Clinical Study
Brief Title: Effects of Kinesio Taping and Extracorporeal Shock Wave Therapy in the Calcaneal Spur
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 26.09.2023 / 4096
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Calcaneal Spur; Plantar Fasciitis; Heel Pain
Keywords: calcaneal spur; extracorporeal shock wave therapy; kinesio taping; plantar fasciitis
MeSH Terms: conditions — Heel Spur; Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : ESWT treatment group: ESWT treatment is applied once a week for 5 weeks
- Group 2 : Kinesio taping treatment group: Kinesio taping was also applied once a week, for a total of 5 sessions. The rake method was used for kinesio taping.

SUMMARY:
The term "heel pain" is used to describe a common, painful condition that is localized in the plantar part of the heel and worsens when weight is placed on the heel. Patients with heel pain are more likely to have thickened plantar fascia, abnormal plantar fascia tissue, thicker plantar heel fat pad, and calcaneal spur. Calcaneal spurs are bony protrusions that typically occur just in front of the medial calcaneal tuberosity. Systemic medical treatments, physical therapy agents, exercise and local injections are often applied for heel pain caused by plantar fasciitis and calcaneal spur.

This study is to examine the effects of ESWT and kinesio taping on pain and other clinical outcomes in patients with calcaneal spurs.

DETAILED DESCRIPTION:
The responses of patients who underwent ESWT or kinesio taping due to calcaneal spur before and after treatment will be compared. Pain, functionality and quality of life are the clinical parameters compared.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over with heel pain
* A calcaneal spur seen on foot radiographs

Exclusion Criteria:

* Those who had received a steroid injection into the heel within the past three months
* Those who had experienced trauma or surgery to the foot and ankle within the past six months
* Those with a rheumatic disease affecting the foot and ankle (e.g., spondyloarthritis)
* Those with open wounds or infections in the area to be treated with lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the Physical Medicine and Rehabilitation outpatient clinic of Şişli Hamidiye Etfal Training and Research Hospital with complaints of heel pain were evaluated. The data of patients who underwent ESWT and kinesio taping were compared with the information on the hospital system.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Pain level before treatment and 3rd month after treatment | From enrollment to the end of treatment at 3rd month
  Pain level will be evaluated with the Numerical Rating Scale. (minimum: 0, maximum: 10)

SECONDARY OUTCOMES:
Assessment of heel sensitivity | From enrollment to the end of treatment at 3rd month
  It will be evaluated with the Heel Tenderness index. (0=no pain; 1=painful; 2=painful and whines; 3=painful, whines, and withdraws)
Assessment of functionality | From enrollment to the end of treatment at 3rd month
  Foot Function Index was used. The FFI consists of 23 items divided into 3 subscales that quantify the impact of foot pathology on pain, disability, and activity limitation in patients. Pain, disability, and activity limitation subscale scores range from 0 to 100.
Assessment of quality of life | From enrollment to the end of treatment at 3rd month
  The 12-item short-form health survey (SF-12) quality of life scale was used to evaluate general quality of life. It was presented as a physical component score (PCS) and mental component score (MCS). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided